CLINICAL TRIAL: NCT02807948
Title: A Clinical Evaluation of the Diagnostic Utility of MRI Scans in Patients Implanted With St. Jude Medical Pacemakers, Implantable Cardioverter Defibrillator, and Cardiac Resynchronization Therapy Devices.
Brief Title: SJM MRI Diagnostic Imaging Registry (IDE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJM-CIP-10130
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Arrhythmia
Keywords: MRI Scan, pacemakers, ICD, CRT
MeSH Terms: conditions — Arrhythmias, Cardiac; Creatine deficiency, X-linked | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pacemaker, ICD, or CRT device patients (Other): Subjects who need a non-thoracic clinically indicated scan
  Interventions: Device: Pacemaker, ICD, or CRT device

INTERVENTIONS:
Device: Pacemaker, ICD, or CRT device — MRI Scans on SJM device implanted subjects for clinical purpose

SUMMARY:
This study is a prospective, non-randomized, multi-center study of subjects implanted with an SJM pacemakers, implantable cardioverter defibrillator (ICD), and cardiac resynchronization therapy (CRT) devices who are clinically indicated for a non-thoracic MRI scan.

DETAILED DESCRIPTION:
This study will be performed as part of a regulated, prospective, non-randomized, multi-center clinical study.

Subjects will be enrolled, undergo a clinically-indicated MRI scan, and have an assessment of adverse events, device measurements, and clinical utility of the MRI scan images.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is implanted with a market-released St. Jude Medical pacemaker, ICD, or CRT current generation device listed in the study protocol and any market-released pacing or defibrillation lead.
2. Patient's device and all leads must be implanted for at least 6 weeks prior to the scheduled date of the MRI.
3. Patient has a clinical indication for a non-thoracic MRI scan, where MRI is the imaging modality of choice that will give adequate results to manage the patient.
4. Patient is scheduled for a non-thoracic MRI scan up to 1.5T.
5. Patient has a pacemaker, ICD, or CRT device implanted pectorally.
6. Patient has the ability to provide informed consent for study participation and be willing and able to comply with the study procedures.
7. Patient is 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Patient has an ICD/CRT-D and is pacemaker dependent
2. Capture threshold is greater than 2.5 volts at 0.5 ms for RA and RV leads
3. Pacing lead impedance is NOT within range (i.e. ≥ 200 and ≤ 2000 ohms)
4. High voltage lead impedance (HVLI) is NOT within range (i.e. ≥ 20 and ≤ 200 ohms)
5. Patient has a device generator battery voltage at elective replacement interval (ERI)
6. Patient has another existing active implanted medical device (e.g. neurostimulator, infusion pump, etc.) that has MR labeling that will not allow the MRI scans to be completed.
7. Patient has other non-MRI compatible device or material implanted

   NOTE:
   * MRI compatible knee replacements, hip replacements, stents, etc. may be included as long as the labeling of these devices allow MRI scans conducted per this protocol
   * MRI compatible mechanical, prosthetic, and bioprosthetic heart valves may be included as long as the labeling of these devices allow for MRI scans conducted per this protocol
   * Non-removable dental implants may be included
8. Patient has a lead extender, adaptor, or capped/abandoned lead
9. Patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, Study Director — Abbott Medical Devices
Locations (58):
- United States (58):
  - Scottsdale Medical Imaging, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - St. Bernards, Jonesboro, Arkansas
  - Quest Imaging, Bakersfield, California
  - Raymond Schaerf, MD, Burbank, California
  - John Muir Medical Center, Concord, California
  - St. Helena Hospital, Deer Park, California
  - Cardiovascular Consultants Heart Center, Fresno, California
  - Newport Diagnostic Center, Newport Beach, California
  - Pro Health Advance Imaging, North Hollywood, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - St. Mary's Medical Center, San Francisco, California
  - Sansum Clinic - Santa Barbara Medical Foundation, Santa Barbara, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Cardiac Arrhythmia Services, Boca Raton, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Florida Hospital, Orlando, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Community Heart and Vascular, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - King's Daughters Medical Center, Ashland, Kentucky
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Suburban Hospital, Bethesda, Maryland
  - Washington Adventist Hospital, Takoma Park, Maryland
  - McLaren Health Care Corporation, Auburn Hills, Michigan
  - Baptist Medical Center, Jackson, Mississippi
  - Advanced Radiology, Columbia, Missouri
  - St. Luke's Hospital, Kansas City, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri
  - Kearney Regional Medical Center, Kearney, Nebraska
  - Denville Diagnostics and Open MRI LLC, Denville, New Jersey
  - Borg and Ide Imaging, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Novant Clinical Research Institute, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Samaritan Heart & Vascular Institute - Cardiology Dept., Corvallis, Oregon
  - Oregon Medical Group, Eugene, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital - 17th Street, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - East Texas Medical Center, Tyler, Texas
  - Lynchburg General Hospital, Lynchburg, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Swedish Medical Center - Heart & Vascular, Seattle, Washington
  - Aurora Medical Group, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pacemaker or CRT-P Device Patients: Subjects who need a non-thoracic clinically indicated scan
  Pacemaker or Cardiac Re-synchronization Therapy -Pacemaker (CRT-P) device: MRI Scans on SJM device implanted subjects for clinical purpose
- ICD or CRT-D Device Patients: Subjects who need a non-thoracic clinically indicated scan
  Implantable Cardioverter Defibrillatoror (ICD) or a Cardiac Re-synchronization Therapy -Defibrillator (CRT-D) device: MRI Scans on SJM device implanted subjects for clinical purpose
Period: Overall Study
Arm/Group | Pacemaker or CRT-P Device Patients | ICD or CRT-D Device Patients
Started | 132 | 57
Completed | 131 | 57
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pacemaker, ICD, or CRT Device Patients
Number analyzed (Participants) | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 126
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 179
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 174
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 189
Arrhythmia History [Count of Participants; unit: Participants]
  Atrial Arrhythmia | 94
  Ventricular Arrhythmia | 26
  No Arrhythmia History | 69

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of MRI Scans From Pacemakers or CRT-Ps Providing Sufficient Image Quality to Allow for a Diagnostic Interpretation.
Description: Based on the ability of the radiologist to read and provide a diagnosis/report.
Time Frame: 1 month
Population: Proportion of MRI scans from CRT-Ps or Pacemakers providing sufficient image quality for diagnostic interpretation
Measure: Count of Units; unit: MRI Scans
Units Other Than Participants: MRI Scans
Arm/Group | Pacemaker or CRT-P Device Patients
Number analyzed (Participants) | 131
Number analyzed (MRI Scans) | 131
MRI Scans | 129

2. Primary Outcome: The Proportion of MRI Scans From ICDs or CRT-Ds Providing Sufficient Image Quality to Allow for a Diagnostic Interpretation.
Description: Based on the ability of the radiologist to read and provide a diagnosis/report.
Time Frame: 1 month
Population: Proportion of MRI scans from ICDs or CRT-Ds providing sufficient image quality for diagnostic interpretation
Measure: Count of Units; unit: MRI Scans
Units Other Than Participants: MRI Scans
Groups:
- ICD or CRT-D Device Patients: Subjects who need a non-thoracic clinically indicated scan
  Implantable Cardioverter Defibrillator or (ICD) or a Cardiac Re-synchronization Therapy -Defibrillator (CRT-D) device: MRI Scans on SJM device implanted subjects for clinical purpose
Arm/Group | ICD or CRT-D Device Patients
Number analyzed (Participants) | 57
Number analyzed (MRI Scans) | 57
MRI Scans | 56

ADVERSE EVENTS:
Time Frame: Adverse events were collected from study enrollment until 1 month after the MRI scan was performed.
Description: A Clinical Events Committee (CEC) composed of physicians who were not actively involved as investigators in any of the studies under the committee's review, nor may they have any significant financial interest in the technology under study, reviewed and adjudicated all adverse device effects, whether serious or not, and all deaths that were reported during the study.
Arm/Group | Pacemaker, ICD, or CRT Device Patients
All-Cause Mortality (participants affected / at risk) | 1/189
Serious Adverse Events (participants affected / at risk) | 0/189
Other Adverse Events (participants affected / at risk) | 4/189
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacemaker, ICD, or CRT Device Patients (N=189)
Chest Pain/ Discomfort (General disorders) | 2 (2)
Back-Up Operation (Cardiac disorders) | 1 (1) — Device reset going into back up mode
Respiratory Infection (Infections and infestations) | 1 (1) — Respiratory infection reported a few days before MRI scan

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/48/NCT02807948/Prot_SAP_ICF_000.pdf